CLINICAL TRIAL: NCT01377818
Title: Prospective Aleatory Study of Non Invasive Mechanical Ventilation Versus Respiratory Rehabilitation in Hypercapnic Stable Severe COPD
Brief Title: Non Invasive Mechanical Ventilation Versus Respiratory Rehabilitation in Hypercapnic COPD
Acronym: COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Eduardo Márquez martín, Neumología Hospital Virgen del Rocío
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 01/0530; COPD15081978 (Other: HUVRocio)
Record Dates: First submitted 2011-06-16; First posted 2011-06-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2006-03

CONDITIONS: Lung, Hyperlucent; Positive-Pressure Respiration, Intrinsic
Keywords: COPD; Exercise trainig
MeSH Terms: conditions — Lung, Hyperlucent; Positive-Pressure Respiration, Intrinsic; Pulmonary Disease, Chronic Obstructive | interventions — Ventilation; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ventilation (Experimental): Group program of positive pressure ventilation noninvasive
  Interventions: Procedure: ventilation
- exercise training (Experimental): The training program (trained group) was carried out for 12 weeks and sessions of 40 minutes duration:
  d. 20 minutes of bicycle ergometer with an initial charge of about 70% of initial maximal oxygen consumption, increasing the load every two weeks as tolerated.
  e. Weightlifting in 2 sets of 6 replicates of 5 simple exercises. These are held at a station multigimnástica (CLASSIC Fitness Center, KETTLER)
  Interventions: Procedure: excecise training
- exercise training and ventilation (Experimental): Group of exercise training program and noninvasive positive pressure ventilation
  Interventions: Procedure: Both

INTERVENTIONS:
Procedure: ventilation — positive-pressure breathing bilevel (BiPAP ® Respironics, Inc.) Parameters initially programmed be: IPAP 10 cm H2O, EPAP 4 cmH2O, method ST setting yourself respirations 12 breaths minute. The IPAP was progressively increased to a maximum of 20 cm H2O, depending on patient tolerability, clinical response and arterial oxygen saturation was continuously monitored by pulse oximetry, trying to avoid possible leaks through the mask. It can also supply oxygen through a cannula connected to the mask at a flow rate of 2-4 liters per minute to maintain oxygen saturation at around 85-90%.
  Patients aired uninterruptedly during nighttime (minimal between 6-8 hours night).
  Other Names: Non invasive positive ventilation
  Arms: ventilation
Procedure: excecise training — The training program (trained group) was carried out for 12 weeks and sessions of 40 minutes duration:
  * 20 minutes of bicycle ergometer with an initial charge of about 70% of initial maximal oxygen consumption, increasing the load every two weeks as tolerated.
  * Weightlifting in 2 sets of 6 replicates of 5 simple exercises. These are held at a station multigimnástica (CLASSIC Fitness Center, KETTLER)
  Other Names: pulmonary rehabilitation
  Arms: exercise training
Procedure: Both — both types of intervention
  Other Names: ventilation and exercise
  Arms: exercise training and ventilation

SUMMARY:
Objective: To analyze the additional benefits of exercise training application by the non-invasive home mechanical ventilation in patients with stable COPD and hypercapnic respiratory failure. SUBJECT: moderate-severe COPD (FEV1 <60%) in chronic respiratory failure (hypoxemia and hypercapnia PaCO2> 45mmHg). GROUPS: 45 patients included prospectively and randomly into 3 groups of 15: a) training + NIPPV group, b) Group training, c) Group NIPPV. Hypothesis: A training program to the effort associated with treatment with NIPPV significantly increase the effects compared with each treatment. MAIN OBJETIVE: Effects on exercise capacity as measured by the test of endurance cycling and test 6-minute walk (distance). SECONDARY OBJECTIVES: Impact on quality of life and dyspnea, as measured by questionnaire and CRQ, systemic inflammatory response (CRP, IL-8, TNF-α), changes in peripheral muscle strength (1RM test, isometric) and effects score BODE index.

DETAILED DESCRIPTION:
1. POPULATION: Patients with COPD diagnosed according to criteria established by the ATS (American Thoracic Society) and the SEPAR (Spanish Society of Pneumology and Thoracic Surgery) to submit a modereda-severe obstruction to airflow (FEV1 <60%) and a clinical impact of their disease. Patients must have chronic respiratory failure with hypoxemia and hypercapnia (PaCO2> 45 mmHg). Patients should be stable and appropriate therapy.
2. SAMPLE: 45 patients diagnosed at the Department of Pulmonology, Hospital Virgen del Rocío de Sevilla, informed consent.
3. EXCLUSION CRITERIA a. Other cardiorespiratory diseases. b. Systemic diseases c. Disability or discomfort to participate in an exercise program or noninvasive ventilation
4. STUDY GROUP: The patients were prospectively included and randomized to one of three groups of 15 patients:

   * Group exercise training program of positive pressure ventilation and noninvasive.
   * Group exercise training program.
   * Group program Ventilation Noninvasive positive pressure.
5. Variables: All patients underwent the following baseline tests:

   • CXR, elementary analysis, 12-lead electrocardiogram

   • simple spirometry and bronchodilator test

   • Blood gases
   * static lung volumes (FRC, RV, TLC) by plethysmography.
   * Study of diffusion (DLCO) by single breath technique
   * maximum muscle pressures both inspiratory and expiratory.
   * Estimation of muscle strength:

     a. Repetition maximum test (Test 1 RM) b. Maximum isometric quadriceps strength and biceps measured with dynamometer (MIE Myometer ltd. With CAS software) c. Determination of muscular fatigue in the isometric tests of quadriceps and biceps, with the same system dynamometer (MIE Myometer ltd., Software CAS)
   * Stress Test:

     a. Maximum, with cycle ergometer and methodology already known, including: Determining, from the respiratory gases, oxygen consumption, carbon production and indirect anaerobic threshold, breathing pattern (minute ventilation, tidal volume, respiratory rate) , electrocardiography and pulse oximetry during exercise with heart rate control, blood pressure and dyspnea Borg scale.

     b. Submaximal cycle ergometer resistance with 70% of the load reached the ultimate test, with essentially control the resistance time, distance walked, and control of saturation (pulse oximetry) and heart rate achieved.

     c. Shuttle walking test, walk test is performed continuously walk between two points separated 10 meters and control the pace of a hearing.
   * Assessment of dyspnea and quality of life:

     1. Baseline dyspnea index and index of transitional measures functional impairment, magnitude of the task and the magnitude of effort (Test of Mahler).
     2. Assessment of quality of life based on the specific questionnaire (CRQ) proposed by Guyatt for COPD patients and modified for your understanding in Spanish-speaking subjects.
6. STUDY DESIGN:

The training program (trained group) was carried out for 12 weeks and sessions of 40 minutes duration:

1. 20 minutes of bicycle ergometer with an initial charge of about 70% of initial maximal oxygen consumption, increasing the load every two weeks as tolerated.
2. Weightlifting in 2 sets of 6 replicates of 5 simple exercises. These are held at a station multigimnástica (CLASSIC Fitness Center, KETTLER) and are:

   1. Simple bending of the arms (pull cable to the chest "Chest pulls"): effects on the latissimus dorsi, deltoids and biceps. Procedure: Sitting in the face of the tower of strength, approaching the bar to the chest and arm span later after return to the starting position.
   2. Simple extension of the arms (force to the neck "Neck press / shoulder press): Effects on the deltoids and triceps. Procedure: Sitting upright on the bench and held the weight to shoulder height, arm span will be held over his head, slowly returning after bending arms to starting position.
   3. Arm flexion and extension against resistance (Butterfly "Butterfly"): Effects on the pectoral and deltoid muscles. Sitting upright on the bench with your forearms and elbows on a lever, takes it to the midline, giving way slowly to the starting position.
   4. Leg extensions ("Leg extension"): Effects on quadriceps. Sitting on the bench leg extension is performed against resistance.
   5. Leg Curl ("Leg curls): Effects on femoral biceps and calves. Lying prone on the bench legs are flexed against the weight.

      Resistance is increased gradually from 50% of the maximum weight you can lift the patient on one occasion, early in the week, up to 85%. Every two weeks the weight limit is reassessed to adjust the training load in each patient (Test 1 RM).

      The groups that come under the non-invasive ventilation program will do so for 12 weeks. Noninvasive ventilation was initiated with support pressure applied with a bilevel positive pressure ventilator (BiPAP ® Respironics, Inc.) This is a ventilatory support system that maintains pressure at two different levels, a level of positive expiratory pressure, or EPAP ( equivalent to conventional mechanical ventilation PEEP) and a positive inspiratory pressure (IPAP, equivalent to pressure support), even in the presence of flow variations.

      The device can be programmed in different modes. In the spontaneous (S), the system cycles to EPAP to IPAP when the patient's inspiratory flow exceeds 40 ml / sec. over 30 msec. IPAP level is maintained for more than 180 milliseconds and cycles to EPAP when inspiratory flow falls below a certain level, when it detects an expiratory effort or the IPAP is held for more than 3 seconds. Thus, the patient retains control over the respiratory rate, inspiratory flow and time. T mode, the system provides the patient ventilatory support to a programmable frequency without detecting any inspiratory effort (similar to a controlled manner in the conventional mechanical ventilation). ST mode would be intermediate between them and equivalent to assist-control ventilation in a volume ventilator.

      The NIV will be implemented initially through a nasal mask (Respironics) with a size appropriate to the patient, fixed by elastic belts fastened with Velcro, and with sufficient strength to prevent escape but while avoiding excessive pressure in order to achieve maximum comfort the patient. If leaks are important in the mouth that hindered the NIV, is replaced by an oronasal mask (Respironics).

      The first set parameters are: IPAP 10 cm H2O, EPAP 4 cm H2O, and ST mode, setting a respiratory rate of 12 breaths per minute. The IPAP was progressively increased to a maximum of 20 cm H2O, depending on patient tolerability, clinical response and arterial oxygen saturation by pulse oximetry continuously monitored, trying to avoid possible leaks through the mask.It can also supply oxygen through a tube connected to the mask at a rate of 2-4 liters per minute in order to maintain oxygen saturation at around 85-90%.

      Patients were ventilated continuously during the night hours (minimum between 6-8 hours per night).

      Upon completion of 12 weeks of treatment applied according to each study group, all tests were repeated at baseline and compared the results.

   7. EXIT CRITERIA STUDY:
   * Offset of the patient.
   * Loss of 3 or 5 consecutive sessions staple.
   * On the initiative of the patient.

     8. Statistical analysis:

   Analyzing the effect size at the expense of an improvement in work reached about 15 W higher than the stress test, assuming a standard deviation of this parameter of + / - 10W, An alpha of 0.05 and a beta of 0, 1 (statistical power 90%) and calculating a loss ratio of 15%, we estimate a sample size of 15 patients for each group.

   Comparing before and after the training response in each group were performed using a paired t test. Comparisons between groups were made using analysis of variance (ANOVA). The Pearson correlation coefficient and linear regression analysis will allow to examine relationships between physiological variables. Be considered significant at p <0.05. The dispersion of a mean value is expressed as mean + / - standard deviation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with COPD (Chronic Obstructive Pulmonary Disease)
2. airflow obstruction with an FEV1 <60%
3. clinical stability, at least last 3 months
4. Chronic respiratory failure with hypoxemia and hypercapnia (PaCO2> 45 mmHg)

Exclusion Criteria:

1. Presence of musculoskeletal condition that limits or prevents the completion of the exercises.
2. Presence of heart disease that prevents the physical exercise.
3. Patients with bronchiectasis or other respiratory disorder other than COPD
4. inability or discomfort to participate in the exercise or non-invasive ventilation

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
exercise capacity | baseline and end of follow-up period (15 weeks)
  Our primary objective is to verify the beneficial effect on exercise capacity of an exercise training program combined with treatment of positive pressure ventilation noninvasive against each of them separately, in patients with COPD. The improvement in exercise capacity will be assessed by increased resistance time (submaximal exercise test) and distance (test 6-minute walk)

SECONDARY OUTCOMES:
Peripheral muscle strength | baseline and end of follow-up period (15 weeks)
  As secondary objectives, we compare the contributions of the combined treatment of:
  a. Peripheral muscle strength (1RM test, maximal isometric strength by dynamometer) and exchange of gases (ABG)
quality of life | baseline and end of follow-up period (15 weeks)
  Impact on symptoms and quality of life (RCMH, CRQ)
inflammation | baseline and end of follow-up period (15 weeks)
  Control of the systemic inflammatory response through: CRP, IL-8 and TNF-α
BODE | baseline and end of follow-up period (15 weeks)
  BODE index as a sensitive parameter of response to therapeutic intervention in these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Marquez, MD, Principal Investigator — Hospital Universitario Virgen del Rocio